CLINICAL TRIAL: NCT00226642
Title: Behandlung Von Leichten Und Unterschwelligen Depressionen. Eine Randomisierte, Kontrollierte Studie Zum Wirksamkeitsnachweis Eines Serotonin-Wiederaufnahme-Hemmers (SSRI), Einer Kognitiven Verhaltenstherapie Und Einer Freien Therapiewahl ("Treatment of Mild and Subthreshold Depressive Disorders". A Randomized, Controlled Trial on the Efficacy of a Serotonin-Reuptake-Inhibitor (SSRI), a Cognitive-Behavioral Therapy and of Free Choice Between SSRI and CBT")
Brief Title: Treatment of Mild and Subthreshold Depressive Disorders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KNDS-2.1
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2005-09-27 (Estimated); Status verified 2002-02

CONDITIONS: Depression
Keywords: depression; primary care
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Sertralin
Behavioral: Cognitive-behavioral therapy
Drug: Placebo
Behavioral: Non-specific supporting group therapy

SUMMARY:
The purpose of this study is to determine the efficacy of a SSRI, cognitive-bahavioral-therapy and a free choice between SSRI and CBT in a sample of primary care patients suffering from mild to moderate depression.

Hypotheses:

* SSRI is superior to placebo
* CBT is superior to a non-specific supporting group therapy

ELIGIBILITY:
Inclusion Criteria:(e.g.)

* subthreshold and mild depressive disorders including dysthymia (HAMD: 8-22)
* informed consent
* 18 years

Exclusion Criteria:(e.g.)

* severe mood disorders
* bipolar disorder
* recurrent brief depression
* suicidality
* alcohol or drug dependency
* obsessive-compulsive disorder
* schizoaffective disorder / schizophrenia
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369

PRIMARY OUTCOMES:
HAMD (changes between baseline and individual endpoint)
IDS (changes between baseline and individual endpoint)

SECONDARY OUTCOMES:
BDI (changes between baseline and individual endpoint)
CGI (changes between baseline and individual endpoint)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Hegerl, Prof, MD, Principal Investigator — LMU, Department of Psychiatry
Locations (1):
- Ludwig-Maximilians-University, Department of Psychiatry, Munich, Germany

REFERENCES:
- [Derived] Mergl R, Allgaier AK, Hautzinger M, Coyne JC, Hegerl U, Henkel V. One-year follow-up of a randomized controlled trial of sertraline and cognitive behavior group therapy in depressed primary care patients (MIND study). J Affect Disord. 2018 Apr 1;230:15-21. doi: 10.1016/j.jad.2017.12.084. Epub 2018 Jan 2. PMID 29355727
- [Derived] Helmreich I, Wagner S, Mergl R, Allgaier AK, Hautzinger M, Henkel V, Hegerl U, Tadic A. Sensitivity to changes during antidepressant treatment: a comparison of unidimensional subscales of the Inventory of Depressive Symptomatology (IDS-C) and the Hamilton Depression Rating Scale (HAMD) in patients with mild major, minor or subsyndromal depression. Eur Arch Psychiatry Clin Neurosci. 2012 Jun;262(4):291-304. doi: 10.1007/s00406-011-0263-x. Epub 2011 Sep 30. PMID 21959915
- [Derived] Mergl R, Henkel V, Allgaier AK, Kramer D, Hautzinger M, Kohnen R, Coyne J, Hegerl U. Are treatment preferences relevant in response to serotonergic antidepressants and cognitive-behavioral therapy in depressed primary care patients? Results from a randomized controlled trial including a patients' choice arm. Psychother Psychosom. 2011;80(1):39-47. doi: 10.1159/000318772. Epub 2010 Oct 23. PMID 20975325
- [Derived] Hegerl U, Hautzinger M, Mergl R, Kohnen R, Schutze M, Scheunemann W, Allgaier AK, Coyne J, Henkel V. Effects of pharmacotherapy and psychotherapy in depressed primary-care patients: a randomized, controlled trial including a patients' choice arm. Int J Neuropsychopharmacol. 2010 Feb;13(1):31-44. doi: 10.1017/S1461145709000224. Epub 2009 Apr 3. PMID 19341510